### Sun-safe Habits Intervention and Education

### NCT04341064

Last approval date: 6/1/2024

Combined for Clinical Trials: 1/10/2025



## SHINE (Sun-safe Habits Intervention and Education) Parental Permission Document

#### STUDY SUMMARY

We invite your child to take part in SHINE because they are a high school student in Utah. It is you and your child's choice whether to participate.

The purpose of the study is to provide skin cancer prevention education in Utah schools. We are doing this study because Utah has the highest rate of melanoma in the U.S. The study will last approximately sixteen months. Everyone in the study will be asked to answer questionnaires and receive information about skin cancer risk factors and prevention strategies.

There are minimal foreseeable risks associated with participation in this project. Participation may help your child become more aware of sun protection and skin cancer prevention.

Please take your time and read this information carefully. You should ask the research staff if you have any questions about this study, or if there is anything you do not understand. If you and your child decide they will **NOT** take part in the program, you will be asked to notify the research staff and/or school.

#### STUDY BACKGROUND AND PURPOSE

The purpose of this research study is to provide skin cancer prevention education in Utah schools. Melanoma is the deadliest form of skin cancer. Our goal is to help children and teenagers establish healthy skin cancer prevention habits from a young age.

Before you decide if you want your child to participate in this research project, it is important for you to understand what will be asked of your child. Please read the following information carefully. Ask us if there is anything that is not clear or if you would like more information. Take time to decide whether you will allow your child to take part in this project.

#### STUDY PROCEDURES

We will provide a skin cancer education program to your child and other students at the school. Your child's school will be randomly assigned to receive either SHINE or a standardized skin cancer education program. What group a school is in will be decided by chance, like flipping a coin.

Both programs will include education on sun protection and skin cancer prevention. Additional parts of the SHINE program may include: 1) interactive activities to illustrate these concepts and help your child plan to do skin cancer prevention behaviors, 2) your child's face being photographed using a camera that shows skin damage from ultraviolet radiation (UVR) exposure, and 3) your child being asked to wear a device (similar to a fitness tracker) that records your child's UVR exposure, and 4) your child being asked to complete daily questionnaires about their outdoor activities during the time they are wearing the UVR exposure device.



Students in both groups will be asked to complete a baseline questionnaire before the program, and a total of up to four follow-up assessments: two short-term assessments one month after the program and the summer following the program, and two longer-term assessments one year after the baseline questionnaire and one year after the program sessions. After the final assessment, your child may be asked to provide additional feedback on the program through a questionnaire and/or interview.

Our study procedures include text messages, phone calls, and emails from the SHINE study to study participants to distribute study assessments.

#### **RISKS**

Although unlikely, it is possible that participation in this study could involve the following risks:

Risks associated with UVR photo: Participants may be shown an image of their face taken with a UV camera. They might see skin damage caused by the sun or other sources (e.g., sunburn, aging, mole excision scars). Some participants may be uncomfortable or concerned about indications of sun damage that may show up in the pictures.

Risks associated with answering study questions: There is minimal risk associated with answering the study questions. Participants do not have to answer any questions that they do not want to answer. They may stop answering questions at any time. All of their answers will remain confidential.

Students who choose to participate in the study will be asked to complete activities (e.g., questionnaires, educational sessions) that take class time. Depending on the school's preferences, the time spent completing study procedures may affect other class activities.

Even though we do everything we can to protect the identity and privacy of participants, there is still a risk that data could be traced back to an individual or family. Some data that have been distributed for approved research use cannot be retrieved.

#### **BENEFITS**

We cannot promise any direct benefit to your child for taking part in this project.

#### **ALTERNATIVE PROCEDURES**

Your child has the option to not be part of this study. You can decide they should stop at any time. The study team will work with your child's school to devise an alternative procedure consistent with the school's instructional methods for students who do not participate in the research study. If you or your child decides that your child will not participate in this study, your child may participate in alternative activities as dictated by your child's school, and your child may also still participate in the program described in this form. Only students who have consented/assented to participate will be asked to complete the questionnaires.

#### **PERSON TO CONTACT**

FOOTER FOR IRB USE ONLY Version: K0218



[August 21st, 2023]


If you have questions, complaints or concerns about this study, you can contact Dr. Yelena Wu and her team. If you think your child may have been injured from being in this study, please call Dr. Wu at (801) 213-6150. Dr. Wu or one of her colleagues can be reached at this number between 8AM-5PM, Monday through Friday.

Institutional Review Board: Contact the Institutional Review Board (IRB) if you have questions regarding your child's rights as a research participant. Also, contact the IRB if you have questions, complaints or concerns which you do not feel you can discuss with the investigator. The University of Utah IRB may be reached by phone at (801) 581-3655 or by e-mail at irb@hsc.utah.edu.

**Research Participant Advocate:** You may also contact the Research Participant Advocate (RPA) by phone at (801) 581-3803 or by email at <a href="mailto:participant.advocate@hsc.utah.edu">participant.advocate@hsc.utah.edu</a>

#### **VOLUNTARY PARTICIPATION**

It is up to you to decide whether to allow your child to take part in this project. Refusal to allow your child to participate or the decision to withdraw your child from this research will involve no penalty or loss of benefits to which your child is otherwise entitled. This will not affect your child's grade in any way. If you choose to not allow your child to participate, we will work with your child's school and teacher to provide an alternative for the student.

#### RIGHT OF INVESTIGATOR TO WITHDRAW

We expect to continue the study until all participants have been enrolled and all of their information has been collected. However, the study may be stopped at any time by the researchers at this institution. The researcher may also withdraw your child from the study without your approval. One reason this may happen is because the researcher feels it is necessary for your child's health and safety. Another reason is if the entire study is stopped.

#### **COSTS AND COMPENSATION TO PARTICIPANTS**

There will be no cost to you or your child to take part in the research study. All study-related equipment and procedures will be provided at no cost to you or your insurance company.

Students who complete each questionnaire will receive a \$5 gift card after the completion of the assessment questionnaire. Students who complete the summer assessment questionnaire will receive a \$10 gift card after the completion of the summer assessment questionnaire.

Students will be entered into a drawing to receive a \$50 gift card for each questionnaire they complete. Students who complete the follow-up surveys will be entered into a drawing to receive a \$75 gift card. Each student who completes the questionnaires will have an equal chance of being selected to receive the gift card.

Students selected to wear a UV sensor will receive \$2 for every sensor check-in questionnaire they complete, with a \$1 bonus for completing all 7 questionnaires (\$15 total). Students who return their devices will receive \$15.

Students who complete a study feedback interview will receive \$10.



#### **NUMBER OF PARTICIPANTS**

We expect to enroll approximately 10,250 high-school students in Utah.

#### CONFIDENTIALITY

By allowing your child to participate in this study, you allow us, the researchers in this study, and others working with us to use some information about your child for this research study.

This is the information we will use and include in our research records:

- Demographic and identifying information like name, diagnosis, gender, age, race, level of schooling, and information about relatives.
- Related medical information about your child like who in the family has been diagnosed with melanoma or any form of cancer.

#### How we will protect and share your child's information:

- We will do everything we can to keep your child's information confidential but we cannot guarantee this. Study information will be kept in a secured manner and electronic records will be password protected. Study information may be stored in your child's research record but not in their medical record.
- In order to conduct this study and make sure it is conducted as described in this form, the
  research records may be used and reviewed by others who are working with us on this
  research:
  - Members of the research team at University of Utah
  - The University of Utah Institutional Review Board (IRB), which reviews research involving people to make sure the study protects your rights
- If we share your child's identifying information with groups outside of University of Utah Health, they may not be required to follow the same federal privacy laws that we follow. They may also share your child's information again with others not described in this form.
- If you do not want us to use information about your child's health, your child should not be part of this research. If you choose not to allow your child to participate, you can still receive health care services at University of Utah Health.

### What if I decide to not allow my child to participate after I sign the Parental Permission Form?

You can tell us anytime that you do not want your child to be in this study and do not want us to use your child's personal information. You can also tell us in writing. If you change your mind, we will not be able to collect new personal information about your child, and they will be withdrawn from the research study. However, we can continue to use personal information we have already started to use in our research, as needed to maintain the integrity of the research.

This authorization does not have an expiration date.



#### **PARENTAL PERMISSION**

If you do not want your child to participate in the SHINE study in-school skin cancer prevention and education activities, and/or in the UVR monitoring follow-up, please contact your child's school at: School Contact Information Or the SHINE study team at: Phone: (801) 213-6131 Email: SHINE@hci.utah.edu

If a response is not received from you by \_\_\_\_\_\_, we will enroll your child in the study.





## SHINE (Sun-safe Habits Intervention and Education) Consent Document

#### **STUDY SUMMARY**

[June 27<sup>th</sup>, 2023]

We invite you take part in SHINE because you are a high school student in Utah. It is your choice whether to participate.

The purpose of the study is to provide skin cancer prevention education in Utah schools. We are doing this study because Utah has the highest rate of melanoma in the U.S. The study will last approximately sixteen months. Everyone in the study will be asked to answer questionnaires and receive information about skin cancer risk factors and prevention strategies.

There are minimal foreseeable risks associated with participation in this project. Participation may help you become more aware of sun protection and skin cancer prevention.

Please take your time and read this information carefully. You should ask the research staff if you have any questions about this study, or if there is anything you do not understand. If you decide you will **NOT** take part in the program, you will be asked to notify the research staff and/or school.

#### STUDY BACKGROUND AND PURPOSE

The purpose of this research study is to provide skin cancer prevention education in Utah schools. Melanoma is the deadliest form of skin cancer. Our goal is to help children and teenagers establish healthy skin cancer prevention habits from a young age.

Before you decide if you want to participate in this research project, it is important for you to understand what will be asked of you. Please read the following information carefully. Ask us if there is anything that is not clear or if you would like more information. Take time to decide whether you will take part in this project.

#### STUDY PROCEDURES

We will provide a skin cancer education program to you and other students at the school. Your school will be randomly assigned to receive either SHINE or a standardized skin cancer education program. What group a school is in will be decided by chance, like flipping a coin.

Both programs will include education on sun protection and skin cancer prevention. Additional parts of the SHINE program may include: 1) interactive activities to illustrate these concepts and help you plan to do skin cancer prevention behaviors, 2) your face being photographed using a camera that shows skin damage from ultraviolet radiation (UVR) exposure, 3) you being asked to wear a device (similar to a fitness tracker) that records your UVR exposure, and 4) you being asked to complete daily questionnaires about your outdoor activities during the time you are wearing the UVR exposure device. Location information from the app is collected on a city level (e.g., SLC, UT) and will only be collected if you choose to allow the app to access your location. Students in both groups will be asked to complete a baseline questionnaire before the program, and a total of four follow-up assessments: two short-term assessments one month after the



University of Utah Institutional Review Board Approved 6/30/2023

IRB\_00118620

[Dr. Yelena Wu] 

[SHINE (Sun-safe Habits Intervention and Education)]

[June 27<sup>th</sup>, 2023]

program and the summer following the program, and two longer-term assessments one year after the baseline questionnaire and one year after the program sessions. After the final assessment, you may be asked to provide additional feedback on the program through a questionnaire and/or interview. Our study procedures include text messages, phone calls, and emails from the SHINE study to study participants to distribute study assessments.

#### **RISKS**

Although unlikely, it is possible that participation in this study could involve the following risks: Risks associated with UVR photo: Participants may be shown an image of their face taken with a UV camera. They might see skin damage caused by sun or other sources (e.g., sun burn, aging, mole excision scars). Some participants may be uncomfortable or concerned about indications of sun damage that may show up in the pictures.

Risks associated with answering study questions: There is minimal risk associated with answering the study questions. Participants do not have to answer any questions that they do not want to answer. They may stop answering questions at any time without affecting their medical care. All of their answers will remain confidential.

Students who choose to participate in the study will be asked to complete activities (e.g. questionnaires, educational sessions) that take class time. Depending on the school's preferences, the time spent completing study procedures may affect other class activities.

Even though we do everything we can to protect the identity and privacy of participants, there is still a risk that data could be traced back to an individual or family. Some data that have been distributed for approved research use cannot be retrieved.

#### **BENEFITS**

We cannot promise any direct benefit to you for taking part in this project.

#### **ALTERNATIVE PROCEDURES**

You have the option to not be part of this study. You can decide to stop at any time. The study team will work with your school to devise an alternative procedure consistent with the school's instructional methods for students who do not participate in the research study. If you decides that you will not participate in this study, you may participate in alternative activities as dictated by your school, and you may also still participate in the program described in this form. Only students who have consented/assented to participate will be asked to complete the questionnaires.

#### PERSON TO CONTACT

If you have questions, complaints or concerns about this study, you can contact Dr. Yelena Wu. If you think you may have been injured from being in this study, please call Dr. Wu at (801) 213-6150. Dr. Wu or one of her colleagues can be reached at this number between 8AM-5PM, Monday through Friday.

Institutional Review Board: Contact the Institutional Review Board (IRB) if you have questions regarding your rights as a research participant. Also, contact the IRB if you have questions, complaints or concerns which you do not feel you can discuss with the investigator. The



[Dr. Yelena Wu] 

[SHINE (Sun-safe Habits Intervention and Education)] [June 27<sup>th</sup>, 2023]

University of Utah IRB may be reached by phone at (801) 581-3655 or by e-mail at irb@hsc.utah.edu.

**Research Participant Advocate:** You may also contact the Research Participant Advocate (RPA) by phone at (801) 581-3803 or by email at <a href="mailto:participant.advocate@hsc.utah.edu">participant.advocate@hsc.utah.edu</a>

#### **VOLUNTARY PARTICIPATION**

It is up to you to decide whether to take part in this project. Refusal to participate or the decision to withdraw from this research will involve no penalty or loss of benefits to which you are otherwise entitled. This will not affect your grade in any way. If you choose to participate, we will work with your school and teacher to provide an alternative for you.

#### **RIGHT OF INVESTIGATOR TO WITHDRAW**

We expect to continue the study until all participants have been enrolled and all of their information has been collected. However, the study may be stopped at any time by the researchers at this institution. The researcher may also withdraw you from the study without your approval. One reason this may happen is because the researcher feels it is necessary for your health and safety. Another reason is if the entire study is stopped.

#### COSTS AND COMPENSATION TO PARTICIPANTS

There will be no cost to you to take part in the research study. All study-related equipment and procedures will be provided at no cost to you or your insurance company.

Students who complete each questionnaire will receive a \$5 gift card after the completion of the assessment questionnaire. Students who complete the summer assessment questionnaire will receive a \$10 gift card after the completion of the summer assessment questionnaire.

Students will be entered into a drawing to receive a \$50 gift card for each questionnaire they complete. Students who complete the follow-up surveys will be entered into a drawing to receive a \$75 gift card. Each student who completes the questionnaires will have an equal chance of being selected to receive the gift card.

Students selected to wear a UV sensor will receive \$2 for every sensor check-in questionnaire they complete, with a \$1 bonus for completing all 7 questionnaires (\$15 total). Students who return their devices will receive \$15.

Students who complete a study feedback interview will receive \$10.

#### **NUMBER OF PARTICIPANTS**

We expect to enroll approximately 10,250 high-school students in Utah.




#### CONFIDENTIALITY

Participating in this study means you allow us, the researchers in this study, and others working with us to use some information about you for this research study.

This is the information we will use and include in our research records:

- Demographic and identifying information like name, diagnosis, gender, age, race, level of schooling, and information about relatives.
- Related medical information about you like who in the family has been diagnosed with melanoma or any form of cancer.

#### How we will protect and share your information:

- We will do everything we can to keep your information confidential but we cannot guarantee
  this. Study information will be kept in a secured manner and electronic records will be
  password protected. Study information may be stored in your research record but not in
  your medical record.
- In order to conduct this study and make sure it is conducted as described in this form, the
  research records may be used and reviewed by others who are working with us on this
  research:
  - Members of the research team at University of Utah
  - The University of Utah Institutional Review Board (IRB), which reviews research involving people to make sure the study protects your rights
- If we share your identifying information with groups outside of University of Utah Health, they may not be required to follow the same federal privacy laws that we follow. They may also share your information again with others not described in this form.
- If you do not want us to use information about your health, you should not be part of this research. If you choose not to participate, you can still receive health care services at University of Utah Health.

#### What if I decide to Not Participate later on?

You can tell us anytime that you do not want to be in this study and do not want us to use your personal information. You can also tell us in writing. If you change your mind, we will not be able to collect new personal information about you, and you will be withdrawn from the research study. However, we can continue to use personal information we have already started to use in our research, as needed to maintain the integrity of the research.

This authorization does not have an expiration date.



#### CONSENT

If you **do not** want to participate in the SHINE study **in-school skin cancer prevention and education activities**, and/or in the **UVR monitoring follow-up**, please contact your school at:

| School Contact Information | |
|------------------------------------------------------------|-----------------|
| Or the SHINE Study Team at: | |
| Phone: (801) 213-6131<br>Email: <u>SHINE@hci.utah.edu</u> | |
| If a response is not received from you byyou in the study. | , we will enrol |





#### SHINE (Sun-safe Habits Intervention and Education) Assent/Consent and Parental Permission Document

#### STUDY SUMMARY

[June 27, 2023]

We invite you take part in SHINE because you are a high school student in Utah. It is your choice whether to participate.

The purpose of the study is to provide skin cancer prevention education in Utah schools. We are doing this study because Utah has the highest rate of melanoma in the U.S. The study will last approximately sixteen months. Everyone in the study will be asked to answer questionnaires and receive information about skin cancer risk factors and prevention strategies.

There are minimal foreseeable risks associated with participation in this project. Participation may help you become more aware of sun protection and skin cancer prevention.

Please take your time and read this information carefully. You should ask the research staff if you have any questions about this study, or if there is anything you do not understand. If you decide you will **NOT** take part in the program, you will be asked to notify the research staff and/or school.

#### STUDY BACKGROUND AND PURPOSE

The purpose of this research study is to provide skin cancer prevention education in Utah schools. Melanoma is the deadliest form of skin cancer. Our goal is to help children and teenagers establish healthy skin cancer prevention habits from a young age.

Before you decide if you want to participate in this research project, it is important for you to understand what will be asked of you. Please read the following information carefully. Ask us if there is anything that is not clear or if you would like more information. Take time to decide whether you will take part in this project.

#### STUDY PROCEDURES

We will provide a skin cancer education program to you and other students at the school. Your school will be randomly assigned to receive either SHINE or a standardized skin cancer education program. What group a school is in will be decided by chance, like flipping a coin.

Both programs will include education on sun protection and skin cancer prevention. Additional parts of the SHINE program may include: 1) interactive activities to illustrate these concepts and help you plan to do skin cancer prevention behaviors, 2) your face being photographed using a camera that shows skin damage from ultraviolet radiation (UVR) exposure, and 3) you being asked to wear a device (similar to a fitness tracker) that records your UVR exposure, and 4) you being asked to complete daily questionnaires about your outdoor activities during the time you are wearing the UVR exposure device. Location information from the app is collected on a city level (e.g., SLC, UT) and will only be collected if you choose to allow the app to access your location. Students in both groups will be asked to complete a baseline questionnaire before the program, and a total of four follow-up assessments: two short-term assessments one month after the program and the summer following the program, and two longer-term assessments one year after the baseline questionnaire and one year after the program sessions. After the final

FOOTER FOR IRB USE ONLY Version: K0218



[Dr. Yelena Wu]
[SHINE (Sun-safe Habits Intervention and Education)]


assessment, you may be asked to provide additional feedback on the program through a questionnaire and/or interview. At the conclusion of the study, data will not be returned to participants with the exception of the UVR photos. Our study procedures include text messages, phone calls, and emails from the SHINE study to study participants to distribute study assessments. By signing this, you are opting into these study communications.

#### **RISKS**

[June 27, 2023]

Although unlikely, it is possible that participation in this study could involve the following risks:

Risks associated with UVR photo: Participants may be shown an image of their face taken with a UV camera. They might see other skin damage caused by the sun or other sources (e.g., sun burn, aging, mole excision scars). Some participants may be uncomfortable or concerned about indications of sun damage that may show up in the pictures.

Risks associated with answering study questions: There is minimal risk associated with answering the study questions. Participants do not have to answer any questions that they do not want to answer. They may stop answering questions at any time without affecting their medical care. All of their answers will remain confidential.

Students who choose to participate in the study will be asked to complete activities (e.g., questionnaires, educational sessions) that take class time. Depending on the school's preferences, the time spent completing study procedures may affect other class activities.

Even though we do everything we can to protect the identity and privacy of participants, there is still a risk that data could be traced back to an individual or family. Some data that have been distributed for approved research use cannot be retrieved.

#### **BENEFITS**

We cannot promise any direct benefit to you for taking part in this project.

#### **ALTERNATIVE PROCEDURES**

You have the option not be part of this study. You can decide to stop at any time. The study team will work with your school to devise an alternative procedure consistent with the school's instructional methods for students who do not participate in the research study. If you decide that you will not participate in this study, you may participate in alternative activities as dictated by your school, and you may also still participate in the program described in this form. Only students who have consented/assented to participate will be asked to complete the questionnaires.

#### PERSON TO CONTACT

If you have questions, complaints or concerns about this study, you can contact Dr. Yelena Wu. If you think you may have been injured from being in this study, please call Dr. Wu at (801) 213-6150. Dr. Wu or one of her colleagues can be reached at this number between 8AM-5PM, Monday through Friday.





[Dr. Yelena Wu] 

[SHINE (Sun-safe Habits Intervention and Education)]

[June 27, 2023]

Institutional Review Board: Contact the Institutional Review Board (IRB) if you have questions regarding your rights as a research participant. Also, contact the IRB if you have questions, complaints or concerns which you do not feel you can discuss with the investigator. The University of Utah IRB may be reached by phone at (801) 581-3655 or by e-mail at irb@hsc.utah.edu.

Research Participant Advocate: You may also contact the Research Participant Advocate (RPA) by phone at (801) 581-3803 or by email at participant.advocate@hsc.utah.edu

#### **VOLUNTARY PARTICIPATION**

It is up to you to decide whether to take part in this project. Refusal to participate or the decision to withdraw from this research will involve no penalty or loss of benefits to which you are otherwise entitled. This will not affect your grade in any way. If you choose not to participate, we will work with your school and teacher to provide an alternative for you.

#### RIGHT OF INVESTIGATOR TO WITHDRAW

We expect to continue the study until all participants have been enrolled and all of their information has been collected. However, the study may be stopped at any time by the researchers at this institution. The researcher may also withdraw you from the study without your approval. One reason this may happen is because the researcher feels it is necessary for your health and safety. Another reason is if the entire study is stopped.

#### **COSTS AND COMPENSATION TO PARTICIPANTS**

There will be no cost to you to take part in the research study. All study-related equipment and procedures will be provided at no cost to you or your insurance company.

Students who complete each questionnaire will receive a \$5 gift card after the completion of the assessment questionnaire. Students who complete the summer assessment questionnaire will receive a \$10 gift card after the completion of the summer assessment questionnaire.

Students will be entered into a drawing to receive a \$50 gift card for each guestionnaire they complete. Students who complete the follow-up surveys will be entered into a drawing to receive a \$75 gift card. Each student who completes the questionnaires will have an equal chance of being selected to receive the gift card.

Students selected to wear a UV sensor will receive \$2 for every sensor check-in questionnaire they complete, with a \$1 bonus for completing all 7 questionnaires (\$15 total). Students who return their devices will receive \$15.

Students who complete a study feedback interview will receive \$10.

#### **NUMBER OF PARTICIPANTS**

We expect to enroll approximately 10,250 high-school students in Utah.

#### CONFIDENTIALITY

FOOTER FOR IRB USE ONLY Version: K0218



University of Utah Institutional Review Board Approved 6/30/2023

IRB 00118620

[Dr. Yelena Wu]
[SHINE (Sun-safe Habits Intervention and Education)]

[June 27, 2023]

Participating in this study means you allow us, the researchers in this study, and others working with us to use some information about you for this research study.

This is the information we will use and include in our research records:

- Demographic and identifying information like name, diagnosis, gender, age, race, level of schooling, and information about relatives.
- Related medical information about you like who in the family has been diagnosed with melanoma or any form of cancer.

#### How we will protect and share your information:

- We will do everything we can to keep your information confidential but we cannot guarantee this. Study information (e.g., UVR photo, questionnaire data, information obtained from the mobile app) will be kept on secure password protected computers and servers, including UBox, maintained by the Huntsman Cancer Institute and University of Utah. Only research staff will have access to the information obtained for this study. Study information may be stored in your research record but not in your medical record. Stored study data will be used to analyze and summarize the effectiveness of the programs provided. Results obtained from the study will be used in publications and presentations so that other schools and researchers can learn about the effect of the programs for skin cancer prevention.
- In order to conduct this study and make sure it is conducted as described in this form, the research records may be used and reviewed by others who are working with us on this research:
  - o Members of the research team at University of Utah
  - The University of Utah Institutional Review Board (IRB), which reviews research involving people to make sure the study protects your rights
- If we share your identifying information with groups outside of University of Utah Health, they may not be required to follow the same federal privacy laws that we follow. They may also share your information again with others not described in this form.
- If you do not want us to use information about your health, you should not be part of this
  research. If you choose not to participate, you can still receive health care services at University
  of Utah Health.

#### What if I decide to Not Participate later on?

You can tell us anytime that you do not want to be in this study and do not want us to use your personal information. You can also tell us in writing. If you change your mind, we will not be able to collect new personal information about you, and you will be withdrawn from the research study. However, we can continue to use personal information we have already started to use in our research, as needed to maintain the integrity of the research.

This authorization does not have an expiration date.

#### ASSENT/CONSENT AND PARENTAL PERMISSION

FOOTER FOR IRB USE ONLY Version: K0218



University of Utah Institutional Review Board Approved 6/30/2023


| [Dr. Yelena Wu] [SHINE (Sun-safe Habits Intervention and Education)] [June 27, 2023] | |
|---|---|
| I confirm that I have read this consent and auth to ask questions. I agree to take part/allow my cauthorize you to use and disclose health inform explained in this document. | |
| Name of Student | Date |
| Signature of Student | _ |
| Name of Parent | <br>Date |



Signature of Parent

# Consent Cover Letter SHINE Study Interviews/Surveys

Parents, School Staff, Principals, Vice Principals, and District/County Staff

#### **Consent Cover Letter** SHINE Study Interviews/Surveys

The purpose of the SHINE research study is to promote sun safety in Utah schools by providing information about sun protection and skin cancer risk to high school students, parents, teachers, and staff. We are hoping to interview parents, school staff, principals, vice principals, and district/county staff to gather their feedback on the SHINE study and ways that SHINE might be delivered in the future.

By completing this 15-30-minute interview and/or survey, you are consenting to participate in this study. You may be asked questions about your demographic information (e.g., your gender), your connections within the community, personal sun protection history, and viewpoints about SHINE and other sun-safety programs. If you complete this interview/survey, you will receive a \$10 gift card. Also, you may be invited to participate in further follow-up interviews and/or follow up questions.

This study will ask about demographic and identifying information like name and contact information. To do our best in keeping your information confidential, interview /survey data will be stored on password-protected computers and servers, including UBox, maintained by the Huntsman Cancer Institute and University of Utah and Qualtrics. Interviews will be stored as digital audio or video files. A pseudonym will be attached to the interview transcripts. You will not be identified in any publications. The information collected in this research may be used for future research studies.

Your participation is completely voluntary. You may choose not to answer any question and are free to withdraw consent and discontinue participation in this interview at any time for any reason without penalty or loss of benefits.

There are no known risks associated with participating in this study.

If you have any questions complaints or if you feel you have been harmed by this research, please contact Dr. Yelena Wu, University of Utah Huntsman Cancer Institute, at (801) 683-9117.

Contact the Institutional Review Board (IRB) if you have questions regarding your rights as a research participant. Also, contact the IRB if you have questions, complaints or concerns which you do not feel you can discuss with the investigator. The University of Utah IRB may be reached by phone at (801) 581-3655 or by e-mail at irb@hsc.utah.edu.

Research Participant Advocate: You may also contact the Research Participant Advocate (RPA) by phone at (801) 581-3803 or by email at participant.advocate@hsc.utah.edu.

By participating in this interview/survey, you are giving consent to participate in this research and to be audio or video recorded. Thank you for your willingness to participate!



# Passive Consent Study Memo for Students

Student Interview

# SHINE (Sun-safe Habits Intervention and Education) Study Memo Document

Hello!

We greatly appreciate your participation in the SHINE study.

You are receiving this letter to inform you that you have been selected to participate in an interview about your experience as a SHINE participant. This interview will be conducted over zoom or via phone and will take about 10-15 minutes. You will be asked questions about your experience with the study team and to provide feedback on the intervention. You will receive an extra \$10 Amazon e-gift card for participating in the interview.

Please know you have the option not to participate in this interview.

If you do not want to be interviewed, please check the box below within one week:

| I DO NOT want to participate in a SHINE study interview. | |
|----------------------------------------------------------|------|
| Name | Date |
| Sincerely, | |

Jacey Jones SHINE Study Coordinator jacey.jones@hci.utah.edu

Nic Siniscalchi
SHINE Clinical Research Coordinator
801-683-9117
SHINE@HCI.utah.edu



### Passive Consent Study Memo for Parents

Student Interview

# SHINE (Sun-safe Habits Intervention and Education) Study Memo Document

Hello SHINE participant parent or guardian!

We greatly appreciate your student's participation in the SHINE study.

You are receiving this letter to inform you that your student has been selected to participate in an interview about their experience as a SHINE participant. This interview will be conducted over zoom or via phone and will take about 10-15 minutes. They will be asked questions about their experience with the study team and to provide feedback on the intervention. They will receive an extra \$10 Amazon e-gift card for participating in the interview.

Please know you and your student have the option not to participate in this interview.

If you do not want your student to be interviewed, please check the box below within one week:

\_\_\_ I DO NOT want my student to participate in a SHINE study interview.

Student Name

Date

Parent/Guardian Name

Sincerely,

Jacey Jones SHINE Study Coordinator jacey.jones@hci.utah.edu Nic Siniscalchi SHINE Clinical Research Coordinator 801-683-9117 SHINE@HCI.utah.edu



# Active Consent Study Memo for Students

Student Interview

#### **SHINE (Sun-safe Habits Intervention and Education) Study Memo Document**

Hello!

We greatly appreciate your participation in the SHINE study.

You are receiving this letter to inform you that you have been selected to participate in an interview about your experience as a SHINE participant. This interview will be conducted over zoom or via phone and will take about 10-15 minutes. You will be asked questions about your experience with the study team and to provide feedback on the intervention. You will receive an extra \$10 Amazon e-gift card for participating in the interview.

Please know your student have the option not to participate in this interview. If you consent to being interviewed, please sign below.

| Student Name | _ |
|-------------------|------|
| Student Signature | Date |
| Sincerely, | |

**Jacey Jones** SHINE Study Coordinator jacey.jones@hci.utah.edu

Nic Siniscalchi SHINE Clinical Research Coordinator 801-683-9117 SHINE@HCI.utah.edu

**FOOTER FOR IRB USE ONLY** Version: 022012



## Active Consent Study Memo for Parents

Student Interview

# SHINE (Sun-safe Habits Intervention and Education) Study Memo Document

Hello SHINE participant parent or guardian!

We greatly appreciate your student's participation in the SHINE study.

You are receiving this letter to inform you that your student has been selected to participate in an interview about their experience as a SHINE participant. This interview will be conducted over zoom or via phone and will take about 10-15 minutes. They will be asked questions about their experience with the study team and to provide feedback on the intervention. They will receive an extra \$10 Amazon e-gift card for participating in the interview.

Please know you and your student have the option not to participate in this interview. If you consent to your student being interviewed, please sign below.

| Student Name | - |
|---------------------------|---|
| Parent/Guardian Signature | |
| Date: | |
| Sincerely, | |

Jacey Jones SHINE Study Coordinator jacey.jones@hci.utah.edu Nic Siniscalchi SHINE Clinical Research Coordinator 801-683-9117 SHINE@HCI.utah.edu

